CLINICAL TRIAL: NCT05856227
Title: A Multicenter, Open-label, Single-arm, Multiple-dose Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of Ceftobiprole Medocaril in Term and Pre-term Neonates and Infants up to 3 Months of Age With Late-onset Sepsis
Brief Title: Late-onset Sepsis in Term and Pre-term Neonates and Infants up to 3 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPR-PIP-003
Record Dates: First submitted 2023-04-17; First posted 2023-05-12 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Neonatal Sepsis
Keywords: Late-onset sepsis; Neonates; Infants
MeSH Terms: conditions — Neonatal Sepsis | interventions — ceftobiprole medocaril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm: Ceftobiprole (Experimental): Ceftobiprole medocaril: 7.5 mg/kg to 15 mg/kg
  Interventions: Drug: Ceftobiprole medocaril

INTERVENTIONS:
Drug: Ceftobiprole medocaril — Ceftobiprole medocaril: 7.5 mg/kg every 12 hours to 15 mg/kg every 8 hours, administered IV as a 2-hour infusion.

SUMMARY:
This study evaluated the safety, pharmacokinetics and efficacy of ceftobiprole in term and pre-term newborn babies and infants up to 3 months of age with late-onset sepsis (LOS). Ceftobiprole is an antibiotic which belongs to a group of medicines called 'cephalosporin antibiotics'. It is approved for its use to treat adults and children with pneumonia in many European and non-European countries.

DETAILED DESCRIPTION:
This was a multicenter, open-label, single-arm, multiple-dose study of intravenous (IV) ceftobiprole medocaril (prodrug of the active moiety ceftobiprole). It could be combined with ampicillin and/or an aminoglycoside based on the Investigator's judgement according to manufacturer's instructions and/or local standard of care.

Following screening, ceftobiprole was administered as a 2-hour infusion at a dose of 7.5 mg/kg every 12 hours to 15 mg/kg every 8 hours, depending on age and weight.

The target treatment duration was 3-10 days, which could be extended to 14 days if considered clinically necessary by the Investigator.

ELIGIBILITY:
Key Inclusion Criteria:

* Informed consent from parent(s) or other legally acceptable representative (LAR) to participate in the study
* Male or female, with a gestational age of ≥ 24 weeks and a post-natal age ranging from ≥ 3 days to ≤ 3 months
* Diagnosis of documented or presumed bacterial LOS requiring administration of systemic antibiotic treatment
* Sufficient vascular access to receive study drug and to allow blood sampling at a site separate from the study drug infusion line

Key Exclusion Criteria:

* Refractory septic shock not responding to 60 minutes of vasopressor treatment within 48 hours before enrollment
* Proven ventilator-associated pneumonia
* Proven central nervous system infection (e.g., meningitis, brain abscess)
* Proven osteomyelitis, infective endocarditis, or necrotizing enterocolitis
* Impaired renal function or known significant renal disease, as evidenced by an estimated glomerular filtration rate (using the Schwartz formula or other applicable formula) calculated to be less than 2/3 of normal for the applicable age group, OR urinary output < 0.5 mL/kg/h (measured over at least 8 hours), OR requirement for dialysis
* Progressively fatal underlying disease, or life expectancy < 30 days
* Use of systemic antibacterial therapy for longer than 72 hours within 7 days before start of study medication
* Participation in another clinical study with an investigational product within 30 days of enrollment in the current study

Ages: 3 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2023-08-06 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (14):
- United States (2):
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - West Virginia University, Morgantown, West Virginia
- Bulgaria (3):
  - MHAT Dr. Stamen Iliev AD Montana, Neonatology Department, Montana
  - UMHAT "Sveti Georgi" EAD, Pediatric surgery Clinic, Plovdiv
  - "Acibadem City Clinic University Hospital Tokuda" EAD, Neonatology Department, Sofia
- Tallinn Childrens' Hospital, Tallinn, Estonia
- Klinikum der Universität München, Kinderklinik und Kinderpoliklinik im Dr. von Haunerschen Kinderspital, Munich, Bavaria, Germany
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Children Clinical University Hospital - Neonatology Clinic, Riga
- Lithuania (2):
  - Lithuanian Health Science University Hospital Kauno klinikos - Neonatology Clinic, Kaunas
  - Vilnius University Hospital Santaros klinikos - Neonatology Center, Vilnius
- Poland (2):
  - Ginekologiczno-Położniczy Szpital Kliniczny im. Marcinkowskiego, Poznan
  - Szpital Uniwersytecki - Klinika Neonatologii, Wroclaw
- Univerzitna nemocnica Martin, Martin, Slovakia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment was administered in hospital setting
Pre-assignment Details: A total of 11 patients were screened for enrollment in this study, two of whom failed the screening process. Nine patients (six pre-term neonates and three term neonates) were enrolled and assigned to the study treatment
Groups:
- Pre-term Neonates: Pediatric patients (gestational age ≥ 24 to 36 weeks), with post-natal age ranging from ≥ 3 days to ≤ 3 months.
- Term Neonates: Pediatric patients (gestational age ≥ 37 weeks), with post-natal age ranging from ≥ 3 days to ≤ 3 months.
Period: Overall Study
Arm/Group | Pre-term Neonates | Term Neonates
Started | 6 | 3
Completed | 4 | 2
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Due to Investigator absence | 1 | 0
Not completed — Cerebrospinal fluid test positive for S. aureus | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-term Neonates: Pediatric patients (gestational age ≥ 24 to 36 weeks), with post-natal age ranging from ≥ 3 days to ≤ 3 months.
  Patients were treated with ceftobiprole 7.5 mg/kg or 10 mg/kg (bodyweight < 4 kg) infused over 2 hours and administered every 12 hours.
  Ceftobiprole may have been combined with locally-provided ampicillin and/or an aminoglycoside based on the Investigator's judgment.
- Term Neonates: Pediatric patients (gestational age ≥ 37 weeks), with post-natal age ranging from ≥ 3 days to ≤ 3 months.
  Patients were treated with ceftobiprole 10 mg/kg (bodyweight < 4 kg) or 15mg/kg (bodyweight ≥ 4 kg) infused over 2 hours and administered every 12 hours.
  Ceftobiprole may have been combined with locally-provided ampicillin and/or an aminoglycoside based on the Investigator's judgment
- Total: Total of all reporting groups
Arm/Group | Pre-term Neonates | Term Neonates | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: Days] | 19.2 (11.05) | 26.7 (4.51) | 21.7 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 0 | 2
  Poland | 0 | 1 | 1
  Bulgaria | 2 | 1 | 3
  Lithuania | 0 | 1 | 1
  Estonia | 2 | 0 | 2
Gestational age [Mean (Standard Deviation); unit: Weeks] | 28.5 (4.68) | 39.0 (1.73) | 32.0 (6.48)
Baseline weight [Mean (Standard Deviation); unit: gram] | 1429.2 (777.49) | 3156.7 (1094.36) | 2005.0 (1193.01)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs)
Description: Number of patients with AEs, serious adverse events (SAEs), AEs leading to discontinuations and AEs of special interest
Time Frame: Up to 5-7 weeks
Population: The safety population consists of all enrolled patients who received at least one dose of ceftobiprole
Measure: Count of Participants; unit: Participants
Groups:
- Term Neonates: Pediatric patients (gestational age ≥ 37 weeks), with post-natal age ranging from ≥ 3 days to ≤ 3 months.
  Patients were treated with ceftobiprole 10 mg/kg (bodyweight < 4 kg) or 15mg / kg (bodyweight ≥ 4 kg) infused over 2 hours and administered administered every 12 hours. Ceftobiprole may have been combined with locally-provided ampicillin and/or an aminoglycoside based on the Investigator's judgment.
Arm/Group | Pre-term Neonates | Term Neonates
Number analyzed (Participants) | 6 | 3
Participants
  Any AE | 3 | 3
  Study-drug-related AE | 0 | 0
  SAE | 1 | 1
  Study-drug-related SAE | 0 | 0
  AE leading to treatment discontinuation | 0 | 1
  AE of special interest | 1 | 1

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ceftobiprole, Ceftobiprole Medocaril, and Open-ring Metabolite
Description: Observed pharmacokinetic parameter Cmax of ceftobiprole (the active moiety), its pro-drug ceftobiprole medocaril and the open-ring metabolite in term and pre-term neonates with post-natal age up to 3 months
Time Frame: On treatment Day 3 prior to and 2, 4, and 8 hours after the start of the first ceftobiprole infusion of the day
Population: Pharmacokinetics (PK) population All patients who received at least one dose of ceftobiprole and had at least one sample of plasma concentration measurement obtained by the appropriate methodology.
Measure: Median (Full Range); unit: μg/mL
Arm/Group | Pre-term Neonates | Term Neonates
Number analyzed (Participants) | 6 | 3
μg/mL
  Ceftobiprole | 17.2 [11.0 to 22.6] | 28.4 [19.1 to 33.8]
  Ceftobiprole medocaril | 0.585 [0.276 to 5.70] | 0.552 [0.376 to 2.59]
  Open-ring metabolite | 1.18 [0.624 to 1.69] | 1.68 [0.998 to 2.06]

3. Secondary Outcome: Number of Patients With a Clinical Response
Description: Clinical cure rate at the end of treatment (EOT) at day 3-14 and test of cure (TOC) at 7-14 days after last ceftobiprole dose visits in the Intent-to-Treat (ITT) population
Time Frame: Up to 28 days
Population: The ITT population consists of all enrolled patients who received at least one dose of ceftobiprole.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-term Neonates | Term Neonates
Number analyzed (Participants) | 6 | 3
Participants
  EoT: Cure | 4 | 2
  EoT: Failure | 0 | 1
  EoT: Unevaluable | 2 | 0
  TOC: Cure | 4 | 2
  TOC: Failure | 0 | 1
  TOC: Unevaluable | 2 | 0

4. Secondary Outcome: Number of Participants With Improved Signs and Symptoms of Late Onset Sepsis (LOS)
Description: Improved signs and symptoms of LOS (including fever, hypothermia, abnormal heart rate, signs of impaired circulation, petechial rash or sclerema neonatorum, respiratory distress, gastrointestinal distress, irritability, lethargy and/or muscular or arterial hypotonia) assessed at Day 3, EOT, and TOC visits (ITT) populations.
Time Frame: Up to 28 days
Population: The ITT population consists of all enrolled patients who received at least one dose of ceftobiprole.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-term Neonates | Term Neonates
Number analyzed (Participants) | 6 | 3
Participants
  Day 3: Resolved | 1 | 1
  Day 3: Improved | 1 | 0
  Day 3: Unchanged | 3 | 1
  Day 3: Worsened | 0 | 1
  Day 3: Not done | 1 | 0
  EOT: Resolved | 1 | 1
  EOT: Improved | 1 | 0
  EOT: Unchanged | 2 | 1
  EOT: Worsened | 1 | 0
  EOT: Not done | 1 | 1
  TOC: Resolved | 2 | 2
  TOC: Improved | 2 | 0
  TOC: Unchanged | 1 | 0
  TOC: Worsened | 1 | 1
  TOC: Not done | 0 | 0

5. Secondary Outcome: Number of Patients With a Microbiological Response
Description: Microbiological eradication or presumed eradication rate at the EOT and TOC visits.
Time Frame: Up to 28 days
Population: The microbiological Intent-to-treat (mITT) population consists of all patients in the ITT population with a causative pathogen identified at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-term Neonates | Term Neonates
Number analyzed (Participants) | 6 | 3
Participants
  EOT: Eradication | 4 | 1
  EOT: Presumed eradication | 0 | 1
  EOT: Persistence | 0 | 1
  EOT: Unevaluable | 2 | 0
  TOC: Eradication | 4 | 1
  TOC: Presumed eradication | 0 | 1
  TOC: Persistence | 0 | 1
  TOC: Unevaluable | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to 5-7 weeks
Description: Adverse event (AE) collection occurred after first study-drug administration, all AEs are considered to be "treatment emergent".
Arm/Group | Pre-term Neonates | Term Neonates
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/3
Other Adverse Events (participants affected / at risk) | 3/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-term Neonates (N=6) | Term Neonates (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-term Neonates (N=6) | Term Neonates (N=3)
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Intraventricular haemorrhage neonatal (Nervous system disorders) | 1 | 0
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Adrenal haemorrhage (Endocrine disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Sepsis neonatal (Infections and infestations) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1
Oedema (General disorders) | 2 | 0
Withdrawal syndrome (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT05856227/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT05856227/SAP_001.pdf